CLINICAL TRIAL: NCT03473769
Title: Sepsis Pre-Alert Monitoring Intervention: A Phase I Randomized, Single Blind Study to Investigate Targeted Enhanced Monitoring for Sepsis
Brief Title: Sepsis Pre-Alert Monitoring Intervention: Study to Investigate Targeted Enhanced Monitoring for Sepsis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to develop formula for data collection
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: 17-01565
Record Dates: First submitted 2018-03-16; First posted 2018-03-22 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Sepsis
Keywords: Hospital Admission
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vital Signs at 2 Hours + CAM-ICU (Experimental): enhanced vital sign and delirium monitoring in patients for who the per-sepsis algorithm reaches alert threshold.
  Interventions: Other: Vital Signs at 2 Hours; Other: Confusion Assessment method for the ICU (CAM-ICU)
- No Intervention (No Intervention): No intervention. Patient treated per standard of care.

INTERVENTIONS:
Other: Vital Signs at 2 Hours — Patients vital signs assessed at 2 hours of arrival at ICU
  Arms: Vital Signs at 2 Hours + CAM-ICU
Other: Confusion Assessment method for the ICU (CAM-ICU) — patient must have altered mental status/fluctuating course and inattention, and either disorganized thinking or altered level of consciousness to be CAM positive; these features are determined by observing the patient during bedside cognitive testing.
  Arms: Vital Signs at 2 Hours + CAM-ICU

SUMMARY:
Sepsis is a leading cause of death worldwide, and contributes to approximately 750,000 hospitalizations per year, a third of which may die. International guidelines recommend timely interventions, including cultures, fluid resuscitation and antibiotics. Following guideline bundles is associated with a decrease in mortality. Key to timely intervention is timely diagnosis.

Using the Epic sepsis predictive analytic tool, investigators will trigger vital sign and delirium monitoring in patients determined to be at increased risk for developing future sepsis.

The primary objective of this study is to demonstrate reduced mortality in patients for whom the pre-sepsis algorithm threshold is met, and who enhanced monitoring.

DETAILED DESCRIPTION:
A means to identify patients before they become ill may improve the effectiveness of established therapies.Epic's electronic medical record (Epic systems, Verona, WI) contains a surveillance tool that uses predictive analytics to identify patients at risk of becoming septic four hours after the alert becomes active. This affords the opportunity to intervene sooner, but it remains unclear what the best course of action should be in a population at risk of sepsis, only some of which may go on to develop the illness. We propose an automatic intervention, consisting of enhanced monitoring, that is tied to the alert. No therapeutics will be mandated. Instead, additional monitoring information will lead to faster diagnosis and therapy, and improved clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* any inpatient at NYU Langone Health System

Exclusion Criteria:

* not an inpatient at NYU Langone Health System

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Number of in-hospital mortalities | 36 Months

CONTACTS AND LOCATIONS:
Overall Officials: Mark Nunnally, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No